CLINICAL TRIAL: NCT01047956
Title: Evaluation Whether Higher Retention Rate is in Those of Combined Methadone With N-Acetyl-Cysteine Compared to Those With Methadone Alone During a Six-month Study
Brief Title: Compare Methadone Combined With N-Acetyl-Cysteine (NAC) and Methadone Alone for Opioids Astaining
Acronym: MNAC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: C09075
Record Dates: First submitted 2010-01-05; First posted 2010-01-13 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Opioids Use
Keywords: Methadone; NAC; opioids
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MethNAC (Experimental): Methadone and N-acetylcysteine for opioids abstaining
  Interventions: Drug: Methadone; NAC
- Methadone (Active Comparator): Methadone alone
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone; NAC — Methadone NAC
  Arms: MethNAC
Drug: Methadone — Methadone
  Arms: Methadone

SUMMARY:
Evaluation whether higher retention rate is in those of combined methadone with N-Acetyl-Cysteine compared to those with methadone alone during a six-month study.

DETAILED DESCRIPTION:
Material abuse nowadays become a serious public health issue, among these, abusing of opioids is the most serious one. It cause HIV infection rate hiking up, recent years in Taiwan, it impairing people health as well. The successive 2 year methadone substitutive abstaining program makes HIV infection rate remarkable decreasing which proven this public health program is successful in controlling HIV spreading. However, methadone substitutive abstaining program can reduce physically and psychologically dependent with opioids for the opioid abusers, collateral benefit is reducing related criminal behaviors and dangerous contagious behaviors, such as sharing the hyperdermic needle.

On the other hand, using methadone still causes sort of material dependent, for example, part of participants of methadone substitutive abstaining program still keep using heroin, the only change is the amount became lesser, even divert into another illegal drugs, compare before participating this program. In the other word, methadone substitutive abstaining program alleviate the dependence of drug abuser for the drug, but can not cure it once for all. In the pass, some study use methadone and other medicine to eradicate this dependence, still there is no effective way to approach it, it still has long way to go. Previous studies found N-acetylcysteine (NAC), a slimy solvent ingredient in human body, by means of extra-cellular glutamate exchange mechanism, not only maintain glutamate concentration inside the raphe, also alleviate motivation and behavior of addictive patient. From previous reports, N-acetylcysteine could be the silver bullet for the opiods addiction patients. The clinical use of N-acetylcysteine is well established for safety as well as tolerance. N-acetylcysteine is an acetyl-derivative of a human essential amino acid; molecular weight is 163.2, a white crystal chemical. N-acetylcysteine has been used in clinical for years, types are intravenous injection, oral and spray, most of it was used for respiratory related disease, a phlegm reducer, such as chronic obstructive pulmonary disease and cystic fibrosis; besides, N-acetylcysteine can combine with toxic metabolite, acetaminophen, prevent lever necrosis of acetaminophen intoxication, therefore, is an antidote of acetaminophen intoxication. Other than FAD approved for clinical using, N-acetylcysteine seems has other clinical benefits such as illness of kidney from the developer, and can promote functions of central nerve system. N-acetylcysteine also considered as improving cognition amnesia and schizophrenia. Besides, oral N-acetylcysteine usually regards as helping health; it sells in grocery, it also accepted by public as diet supplement. According long term study of oral N-acetylcysteine for patients of chronic obstructive pulmonary disease, only has some minor side-effects, mostly uncomfortable in intestines and stomach, for example, nausea, vomiting and diarrhea. As an antidote of N-acetylcysteine, some cases reported which caused hypertension, chest distress, rectum breeding, respiratory distress, headache, fatigue, fever and rash; those symptoms are intoxication of acetaminophen, it is hard to judge the side-effects came from which one. The side-effects of intravenous N-acetylcysteine include vomiting and diarrhea; some cases indicated 45 (8%) out of 529 patients of acetaminophen intoxication showed allergic reactions, most are skin hypersensitive reaction, such as rash, itch, 18 showed whole-body allergy include, bronchospasm, angioedema and vomiting etc. Those allergies can be alleviated by antihistamine, steroids and adrenalin. Other researchers found patients have 3 fold systemic allergy of asthma history than no history. In general, medicine allergic history will not increase danger of allergic reaction. One case report showed a 2 year old girl, a acetaminophen intoxication patient, caused a serious epilepsy when treated with intravenous injection. Conclude that oral and intravenous of N-acetylcysteine are safe in clinical use, few cases could cause serious side-effects (especially for intravenous type of N-acetylcysteine), and it needs to be careful. From the result of animal test in 2008, gave N-acetylcysteine daily suppressed experimental animal addiction behavior, even still held valid 40 days after stopped injection. Another animal test using male Sprague-Dawley had similar results. According previous results, N-acetylcysteine was used for alleviation of addiction behavior proven in certain effectiveness, if combine with methadone substitutive abstaining program, should increase successful rate. In this study, double-blind prospective study will be used, in methadone substitutive abstaining program to compare N-acetylcysteine is be used or not. This experiment expects methadone come alone with N-acetylcysteine in opioid abstaining will be better results than control group of methadone alone in 6 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-65 years old, all genders.
2. Psychiatry doctor diagnosed who met DSMIV-TR criteria opioid addiction or opioid abusing.
3. Participants need to understand procedures and assays of this experiment.
4. Participants are willing to accept methadone substitutive abstaining program.
5. Participants are willing to provide small amount of blood for testing.
6. Participants are voluntarily to join interview(s), approximately 30-45min.

Exclusion Criteria:

1. Participants have respiratory distress or other respiratory system illnesses.
2. Participants have serious illness and possible die within 1 year or intensive care needed within 6 month.
3. Participants have been diagnosed cardio-vascular disease recently.
4. Participants have allergy to N-acetylcysteine.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD., PhD., Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan